CLINICAL TRIAL: NCT00189202
Title: Efficacy of Sirolimus-Based, Steroid Avoidance Maintenance Immunosuppression in Black de Novo Kidney Transplant Recipients
Brief Title: Efficacy of Sirolimus-Based, Steroid Avoidance Immunosuppression African Americans
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Akinlolu Ojo, Emeritus Professor of Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Steroid Avoidance in A.A.
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-02

CONDITIONS: End Stage Renal Disease; Kidney Transplantation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Sirolimus

ARMS (1):
- Sirolimus, steroid avoidance arm (Experimental): Thymoglobulin induction, sirolimus and no maintenance corticosteroid.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Thymoglobulin induction, sirolimus and no maintenance corticosteroid
  Other Names: Rapamune

SUMMARY:
African Americans receiving a kidney transplant are considered at high risk for early rejection of their transplanted kidney and require more immunosuppression to maintain their kidney transplant function. This increase in immunosuppression puts this group at risk for drug-related toxicities and complications such as post-transplant diabetes.

This study will evaluate:

1. Whether a sirolimus based steroid avoidance regimen in African Americans may decrease the risks of drug-related toxicities,
2. Decreased rates of metabolic complications such as post-transplant diabetes,
3. The effect of Sirolimus plus a reduced dose cyclosporine on renal allograft function.

DETAILED DESCRIPTION:
This is an open labeled prospective trial with race matched historical controls. The treatment group (experimental arm) will be African American de novo solitary renal transplant recipients. The control arm will consist of race matched solitary renal transplant recipients who received a Cyclosporine (CsA) -based immunosuppressive regimen. The subjects will be matched for organ source (living donor vs. cadaveric). The experimental treatment arm will have an immunosuppression regimen consisting of Sirolimus, Reduced dose cyclosporine, Thymoglobulin, and only 3 doses of steroids.

ELIGIBILITY:
Inclusion Criteria:

* African American recipient race
* Solitary cadaveric or living donor renal transplantation
* Age ≥18years at the time of transplantation
* Negative pregnancy serum test in females with childbearing potential

Exclusion Criteria:

* Age < 18 years at the time of transplantation
* Multi-organ transplant recipient
* Currently taking steroids
* White Blood Cell Count < 3,000
* Platelet count < 100,000
* Triglycerides >400mg/dL
* Cholesterol > 350 mg/dL
* Unwillingness to comply with study procedures
* Allergic reaction to sirolimus Allergy to polyclonal antilymphocyte drugs (Thymoglobulin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2004-08; Primary Completion 2008-07-01 (Actual); Study Completion 2008-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akinlolu Ojo, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sirolimus, Steroid Avoidance Arm
Started | 49
Completed | 44
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Population: From the 49 consented, 5 were not begun on treatment or removed very early on for clinical reasons, so they are not included in baseline data.
Arm/Group | Sirolimus, Steroid Avoidance Arm
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Cumulative One-year Acute Rejection Rates
Description: To test the efficacy of Sirolimus (SRL)-based steroid avoidance regimen in high risk de novo renal allograft recipients. Efficacy endpoints for this objective is: cumulative one-year acute rejection rates of the transplant
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus, Steroid Avoidance Arm
Number analyzed (Participants) | 44
Participants | 7
Statistical Analysis 1: Comparison: Sirolimus, Steroid Avoidance Arm; Test type: Equivalence — Equivalence margin 8% plus or minus 4; p = 0.28, Mantel Haenszel

2. Primary Outcome: One-year Graft Survival
Description: To test the efficacy of SRL-based steroid avoidance regimen in high risk de novo renal allograft recipients. Efficacy endpoints for this objective is: one-year graft survival
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus, Steroid Avoidance Arm
Number analyzed (Participants) | 44
Participants | 42
Statistical Analysis 1: Comparison: Sirolimus, Steroid Avoidance Arm; Test type: Other; p = 0.70, Kaplan-Meier

3. Primary Outcome: One-year Patient Survival
Description: To test the efficacy of SRL-based steroid avoidance regimen in high risk de novo renal allograft recipients. Efficacy endpoints for this objective is: one-year patient survival
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus, Steroid Avoidance Arm
Number analyzed (Participants) | 44
Participants | 44

4. Secondary Outcome: Incidence of Post Transplant Diabetes
Description: To determine whether SRL-based steroid avoidance maintenance regimen is associated with decreased rates of metabolic complications. Endpoint is incidence of posttransplant diabetes mellitus
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus, Steroid Avoidance Arm
Number analyzed (Participants) | 44
Participants | 9

5. Secondary Outcome: Drug-treated Dyslipidemic Syndrome
Description: To determine whether SRL-based steroid avoidance maintenance regimen is associated with decreased rates of metabolic complications. Endpoint is drug-treated dyslipidemic syndrome
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus, Steroid Avoidance Arm
Number analyzed (Participants) | 44
Participants | 21

6. Secondary Outcome: Blood Pressure Control
Description: To determine whether SRL-based steroid avoidance maintenance regimen is associated with decreased rates of metabolic complications. Endpoint is number of people who had their blood pressure in the target control range with or without medication
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus, Steroid Avoidance Arm
Number analyzed (Participants) | 44
Participants | 34

ADVERSE EVENTS:
Time Frame: 1 year follow up
Arm/Group | Sirolimus, Steroid Avoidance Arm
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes